CLINICAL TRIAL: NCT05540769
Title: Holter and ECG Changes After Transcatheter Closure Of ASD In Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abdel Galil, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-04-19
Record Dates: First submitted 2022-08-14; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- case group (Experimental)
  Interventions: Procedure: catheter guided ASD closure

INTERVENTIONS:
Procedure: catheter guided ASD closure — transcatheter secundum ASD device closure

SUMMARY:
Atrial septal defects (ASD) account for 10% of all congenital heart defects [1].

Hemodynamic consequences of an ASD are dilatation of the right atrium and right ventricle (RV) because of the volume overload due to the left-to-right shunt through the ASD.For several decades, surgical closure has been considered the standard method of repairing a secundum ASD [2]. Surgical repair, albeit enjoying a high success rate, negligible mortality, and good long-term outcome, is associated with morbidity, discomfort, and thoracotomy scars [3]. That is why the transcatheter closure of the ASD has more recently become an alternative to the surgical procedure [4].

During the last decade , ASD device closure , has finally replaced surgical ASD repair in most patients as the standard method of repair for the secundum ASD[5,6].

Cardiac arrhythmias and right chamber enlargement are well known long-term sequelae of atrial septal defect (ASD) [7]. Therefore, many authors suggest ASD closure before adulthood [8,9].

Classical ECG findings for a significant ASD are prolongation of the PR interval, prolongation of the QRS duration and right axis deviation of the QRS [10].

Percutaneous ASD closure is an ideal situation to study changes of RV dimensions and their impact on ECG as interferences from cardiopulmonary bypass, cardiac incisions and sutures on the right atrium and on the interatrial septum are excluded[11].

DETAILED DESCRIPTION:
The Aim Of Work:

The focus of this study is to describe the electrocardiography (ECG) changes 1,6,12 months after ASD transcatheter device closure in a pediatric population.

Patients and Method:

* Place of the Study: Cardiac catheterization unit , pediatric department , Sohag university hospital .
* Type of the Study: Prospective observational study.
* Study Period: 12 months (starting from the date of obtaining the approval from the research ethics committee) .
* Patients:
* Inclusion Criteria:
* All children under the age of 18 years diagnosed with ASD , that will undergo transcatheter secundum ASD device closure during the period of the study .
* Exclusion Criteria:
* Failure to obtain informed consent .

Ethical consideration Approval will be obtained from the medical research ethics committee (MREC) of faculty of medicine Sohag university .Informed consent will be obtained from parent or authorized legal representative of all children included in the study .

* Methods of the Study:
* The following data will be collected from all patients:

  *Demographic data:
  * Name , Age , sex and Residence .

    *Medical history:
  * General medical history will be obtained .
* All patients will be subjected to :

  * 12 leads ECG (Fukuda Denshi CardiMax ECG device model FCP-7101 with a 25 mm/s paper speed, gain 10 mm/mV) the day before and the day after the procedure
  * Holter ECG (Mortara H3+ Holter ECG) the day before and the day after the procedure.
  * Clinical , ECG and Holter follow-up will be obtained at 1, 6 and 12 months respectively.

Statistical analysis:

The collected data will be statistically analyzed and expressed in tables and charts.

Conclusions and recommendations will be suggested based on the results.

ELIGIBILITY:
Inclusion Criteria:

* - All children under the age of 18 years diagnosed with ASD , that will undergo transcatheter secundum ASD device closure during the period of the study .

Exclusion Criteria:

* - Failure to obtain informed consent .

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
ECG changes in Heart rate [HR] before and after the catheter guided ASD device closure | 1 month , 6 months , 1 year
  12 leads ECG (Fukuda Denshi CardiMax ECG device model FCP-7101 with a 25 mm/s paper speed, gain 10 mm/mV) the day before and the day after the procedure
  -Heart rate [HR]
ECG changes before and after the catheter guided ASD device closure | 1 month , 6 months , 1 year
  12 leads ECG (Fukuda Denshi CardiMax ECG device model FCP-7101 with a 25 mm/s paper speed, gain 10 mm/mV) the day before and the day after the procedure ECG PR interval , ECG QRS interval , ECG axis , and ECG corrected QT interval "QTc" will be recorded .
Holter ECG changes in Heart rate [HR] before and after the ASD closure | 1 month , 6 months , 1 year
  Holter ECG (Mortara H3+ Holter ECG) changes the day before and the day after the procedure.
  Heart rate [HR]
Holter ECG changes before and after the ASD closure | 1 month , 6 months , 1 year
  Holter ECG (Mortara H3+ Holter ECG) changes the day before and the day after the procedure.
  ECG PR interval , ECG QRS interval , ECG axis , and ECG corrected QT interval "QTc" will be recorded .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy JG, Gersh BJ, McGoon MD, Mair DD, Porter CJ, Ilstrup DM, McGoon DC, Puga FJ, Kirklin JW, Danielson GK. Long-term outcome after surgical repair of isolated atrial septal defect. Follow-up at 27 to 32 years. N Engl J Med. 1990 Dec 13;323(24):1645-50. doi: 10.1056/NEJM199012133232401. PMID 2233961
- [Background] Meyer RA, Korfhagen JC, Covitz W, Kaplan S. Long-term follow-up study after closure of secundum atrial septal defect in children: an echocardiographic study. Am J Cardiol. 1982 Jul;50(1):143-8. doi: 10.1016/0002-9149(82)90020-0. PMID 7090997
- [Background] Peters B, Ewert P, Schubert S, Abdul-Khaliq H, Schmitt B, Nagdyman N, Berger F. Self-fabricated fenestrated Amplatzer occluders for transcatheter closure of atrial septal defect in patients with left ventricular restriction: midterm results. Clin Res Cardiol. 2006 Feb;95(2):88-92. doi: 10.1007/s00392-006-0329-3. Epub 2006 Jan 16. PMID 16598516
- [Background] Masura J, Gavora P, Podnar T. Long-term outcome of transcatheter secundum-type atrial septal defect closure using Amplatzer septal occluders. J Am Coll Cardiol. 2005 Feb 15;45(4):505-7. doi: 10.1016/j.jacc.2004.10.066. PMID 15708695